CLINICAL TRIAL: NCT01112527
Title: An Open-Label, Phase 2 Trial of Orally Administered PF-00299804 in Adult Patients With Relapsed/Recurrent Glioblastoma (GBM)
Brief Title: PF-00299804 in Adult Patients With Relapsed/Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Henry Ford Hospital (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Tracy T. Batchelor, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-468; WS573383 (Other: Pfizer); NCT01036477 (obsolete NCT alias)
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Glioblastoma; GBM; Glioblastoma Multiforme
Keywords: PF-00299804
MeSH Terms: conditions — Glioblastoma | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Experimental): Patients with Glioblastoma that has returned or grown after chemotherapy or radiation treatment and who will be having a standard operation to remove the tumor.
  Interventions: Drug: PF-00299804
- Arm B (Experimental): Participants with glioblastoma at first recurrence who are not surgical candidates and who have not had prior anti-VEGF therapy.
  Interventions: Drug: PF-00299804
- Arm C (Experimental): Participants with glioblastoma who are not surgical candidates and who are at first recurrence from a therapeutic regimen containing bevacizumab.
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — Taken orally once a day

SUMMARY:
There are three arms to this study (A, B and C) The purpose of this research study during Arm A is to see how much of PF-00299804 gets into the brain tumor. For many brain tumors, one reason that chemotherapy drugs might not be effective is that the drug may not be able to get into the brain tumor and kill the cancer cells. We will determine how much PF-00299804 gets into the brain tumor by obtaining a sample of the tumor from the surgery that the participant already has scheduled. The purpose of this research study during Arm B and C, is to determine how well PF-00299804 works in killing cancer cells. PF-00299804 works by binding to specific proteins found on the surface of some cancer cells that promote a growth signal. Blocking this signal from reaching its target on the cancer cells may slow or stop the cancer from growing.

DETAILED DESCRIPTION:
ARM A:

* Each treatment cycle lasts four weeks (28 days). There are no breaks from taking PF-00299804 between treatment cycles. Participants will take PF-00299804 once a day for a total of 7 to 9 days before surgery. They will then stop taking PF-00299804 until they have recovered from surgery.
* Once they have recovered from surgery, they will continue to take PF-00299804 once a day until their disease worsens, they experience side effects or they decide to stop study treatment.
* The following tests and procedures will be performed at the time intervals specified: Research blood tests (Day 1 of study drug administration, day of surgery, day 1 of all cycles after surgery, day 14 of the first cycle after surgery); tissue samples (day of surgery); physical and neuro exams (day 1 of all cycles after surgery); skin exam (day 1 of all cycles after surgery and day 14 of the first cycle after surgery).
* An assessment of the tumor by CT or MRI scan will be made within 24 hours after surgery. Another assessment by CT or MRI scan will be made at the end of cycle 2 and then at the end of every even numbered cycle thereafter.

ARM B & C:

* Each treatment cycle lasts four weeks (28 days). There are no breaks from taking PF-00299804 between treatment cycles. Participants will take PF-00299804 orally once a day until their disease worsens, they experience any side effect, or if they decide to stop study treatment.
* Participants will come into the clinic on Day 1 and Day 14 of Cycle 1, and then on Day 1 of all subsequent cycles for some of the following tests and procedures: research blood tests, physical and neuro exams, skin exam, urine test and Patient Reported Outcomes questionnaire.
* An assessment of the participants tumor by CT scan or MRI scans will be done at the end of Cycle 2, 4 and then every other cycle thereafter.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed diagnosis of a recurrent primary WHO grade IV malignant glioma (glioblastoma). Patients with recurrent disease whose diagnostic pathology confirmed glioblastoma will not need re-biopsy. Patients with prior low-grade glioma or anaplastic glioma are eligible if histologic assessment demonstrates transformation to GBM.
* Evidence of EGFR gene amplification by fluorescence in situ hybridization (FISH) in archival tumor material.
* Patients must have at least 15 unstained slides or 1 tissue block (frozen or paraffin embedded) available from a prior biopsy or surgery.
* For Arm A: patients must be at first recurrence of GBM, must not have had previous anti-VEGF therapy, and must be candidates for surgical partial or gross-total resection.
* For Arm B: patients must be at first recurrence of GBM and must not have had prior anti-VEGF therapy.
* For Arm C: patients may have had an unlimited number of prior therapies for GBM, however must be at first recurrence from a therapeutic regimen containing bevacizumab
* Progressive disease on contrast-enhanced brain CT or MRI as defined by McDonald Criteria, or have documented recurrent glioblastoma on diagnostic biopsy.
* Prior to enrollment, there must be an interval of at least 2 weeks between prior surgical resection (1 week for intracranial biopsy) and adequate wound healing.
* Interval of at least 12 weeks from prior radiotherapy unless there is either: a) histopathologic confirmation of recurrent tumor, or b) new enhancement on MRI outside of XRT treatment field.
* Patients must have sufficient time to recover from prior therapy.
* Karnofsky Performance Score 70% or greater
* Adequate hematologic and liver function as outlined in the protocol
* Creatinine within normal institutional limits
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation and for at least 3 months thereafter.

Exclusion Criteria:

* Presence of extra-cranial metastatic disease
* Participants may not be receiving any other investigational agents
* Prior investigational therapy with an agent that is known or proposed to be active by action on any component of the EGFR tyrosine kinase, IGF1R, mTor, orc-MET pathways
* Patients who have been previously treated with an anti-VEGF agent will be excluded from Arm A and Arm B.
* Patients must not have received prior Gliadel wafers
* For participants in Arm A, if the diagnostic pathology of the biopsy specimen is not consistent with recurrent glioblastoma, then the participant must be taken off study and be replaced with another participant that meets the inclusion criteria and is eligible for surgical resection.
* Any surgery (not including minor diagnostic procedures such as lymph node biopsy) within 2 weeks of baseline disease assessments; or not fully recovered from any side effects of previous procedures.
* Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drug.
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this protocol
* Patients with known interstitial lung disease
* Uncontrolled or significant cardiovascular disease
* Any patient with a history of significant cardiovascular disease, even if currently controlled, or who has signs or symptoms suggesting impaired left ventricular function in the judgment of the investigator must have a screening left ventricular ejection fraction evaluation by ECHO or MUGA. Patients with LVEF measurements below local institutional lower limit of normal or less then 50% will not be eligible.
* Individuals with a history of a different malignancy are ineligible except for the circumstances outlined in the protocol
* Patients who have had prior stereotactic radiotherapy, convection enhanced delivery or brachytherapy as gliosis/scarring from these modalities may limit delivery
* Patients will not be eligible if they present with leptomeningeal dissemination
* Pregnant women
* HIV-positive individuals on combination antiretroviral therapy are ineligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PF-00299804
* Other severe acute or chronic medical condition, uncontrolled intercurrent illness or laboratory abnormality that may increase the risk associated with trial participation or investigation product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 2 years
  Assess progression-free survival at six months in patients with recurrent GBM and EGFR amplification in archival tumor material who are treated with continuous daily dosing of PF-00299804 (Arm B)

SECONDARY OUTCOMES:
Ability of PF-00299804 to cross the blood-brain barrier | 2 years
  Assess the ability of PF-00299804 to cross the blood-brain barrier in GBM patients who are candidates for surgical re-section in Arm A.
Safety and tolerability | 2 years
  Evaluate the safety and tolerability of orally administered PF-00299804 on a continuous dosing schedule in patients with recurrent GBM.
Anti-tumor response | 2 years
  Assess anti-tumor response in patients in Arm B

CONTACTS AND LOCATIONS:
Overall Officials: Tracy T. Batchelor, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cleveland Clinic, Cleveland, Ohio